CLINICAL TRIAL: NCT02714075
Title: Comparison of Iron Absorption From Extruded FePP-fortified Rice Containing Different Zinc Compounds, Citric Acid/Trisodium Citrate and Sodium EDTA
Brief Title: Comparison of Iron Absorption From Extruded FePP-fortified Rice Containing Zinc, Citric Acid/Trisodium Citrate and EDTA
Acronym: MM_Rice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University for Development Studies, Tamale, Ghana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MM_Rice
Record Dates: First submitted 2016-03-10; First posted 2016-03-21 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Iron Deficiency and/or Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric pyrophosphate; Zinc Oxide; Zinc Sulfate; Citric Acid; trisodium citrate; Edetic Acid; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iron fortified rice (Experimental): Administration of iron fortified rice to all subjects; subjects will act as their own controls and each subject will receive all foreseen treatments/interventions.
  Interventions: Other: Ferric Pyrophosphate and Zinc Oxide; Other: Ferric Pyrophosphate and Zinc Sulphate; Other: Ferric Pyrophosphate, ZnO, Citric Acid and Trisodium Citrate; Other: Ferric Pyrophosphate, ZnSO4, CA/TSC; Other: Ferric Pyrophosphate, ZnO, CA, EDTA; Other: Ferrous Sulphate

INTERVENTIONS:
Other: Ferric Pyrophosphate and Zinc Oxide — Extruded rice fortified with Ferric Pyrophosphate, Zinc Oxide (ZnO) and micronutrients
Other: Ferric Pyrophosphate and Zinc Sulphate — Extruded rice fortified with Ferric Pyrophosphate, Zinc Sulphate (ZnSO4) and micronutrients
Other: Ferric Pyrophosphate, ZnO, Citric Acid and Trisodium Citrate — Extruded rice fortified with Ferric Pyrophosphate, Zinc Oxide (ZnO), Citric Acid (CA) and Trisodium Citrate (TSC) and micronutrients
Other: Ferric Pyrophosphate, ZnSO4, CA/TSC — Extruded rice fortified with Ferric Pyrophosphate, ZnSO4, CA/TSC and micronutrients
Other: Ferric Pyrophosphate, ZnO, CA, EDTA — Extruded rice fortified with Ferric Pyrophosphate, ZnO, CA, EDTA and micronutrients
Other: Ferrous Sulphate — Extruded rice fortified with micronutrients, Ferrous Sulphate solution will be added at consumption

SUMMARY:
Rice can only be fortified with ferric pyrophosphate (FePP), which is of low bioavailability in human subjects. Compounds such as citric acid/trisodium citrate (CA/TSC) or sodium ethylene-diamine tetraacetic-acid (EDTA) could serve as absorption enhancers. Recent findings from single meal studies indicate CA/TSC to have an enhancing effect on iron absorption from FePP-fortified rice. In contrast, ZnO has been suggested to have detrimental effects. Furthermore, in vitro findings suggest an increased iron solubility from iron and EDTA-co-fortified rice - but the bioavailability in humans remains to be investigated. These effects should thus be investigated in 'real-life' conditions, when fortified rice is implemented in a complete diet administered throughout several days in a target population for a rice fortification program.

Objective: To assess iron absorption from the diet from different iron fortified rice formulations in iron deficient anaemic children.

The investigators aim to conduct an iron absorption study in 30 Ghanaian school-age children investigating different fortification approaches in a multiple meal randomized, cross over study.

DETAILED DESCRIPTION:
Iron of differing molecular weights (54Fe, 56Fe, 57Fe, 58Fe) and other nutrients and additives will be extruded into rice kernels, these kernels will be blended with regular unfortified rice and administered to the study participants.

Recruitment of study participants will be through a local investigator in close collaboration with the Ghanaian school authorities. Before starting the study, 6 children will be asked to participate in a pilot testing, where they will be administered 2 portions of rice (50 g dry weight) with a vegetable sauce with a four hours delay in between the meals. This is to allow the investigators to define, the optimal portion size, that will be used throughout the study. For their participation, the children will receive a small symbolic gift. The investigators envisage screening approximately 60 children living in Tamale and surrounding rural areas at least one week before study start. Recruitment of participants will be done until reaching a number of 30 eligible participants. Participant's caretakers will be explained the study procedures and need to sign a consent form before the participant is exposed to any study procedure. Participants at screening will be assigned a unique study identification (running number and participant's initials), which they will keep if included in the study. All data will be kept confidential. The medical history, dietary intake data and data concerning socioeconomic status will be assessed using questionnaires, body temperature, height and weight will be measured and z-scores (weight for age) will be calculated. A blood sample will be collected from each participant for the initial determination of iron status, detection of parasitic infections (including measurements of hemoglobin (Hb), serum ferritin (SF), soluble transferrin receptor (sTfR), Zinc protoporphyrin to heme ratio (ZPP), C-reactive protein (CRP), Alpha acid glycoprotein, and malaria parasitemia. All screened participants will receive an appropriate dose of an anthelmintic free of charge, unless they had received an according treatment within the last two months. Based on the information obtained from screening, in-/ exclusion criteria will be checked and participant's eligibility will be judged accordingly. Thirty iron deficient and/or anemic children (hereafter called participants) will be included in the absorption study. For the initial determination of the iron status and infection detection, the children will receive a symbolic gift from the investigators. There will be no monetary compensation for participation; however, the children or their caregivers will receive a symbolic gift for completion of the study. Potential transport costs for the children and their caregivers will be covered by the project.

The whole study duration will be eleven weeks (excluding screening and pilot testing). Participants will donate one blood sample at screening and two blood samples during the remaining study period. Between Monday and Friday, the participants will receive two meals per day, one in the morning (first meal) and one at noon (second meal). One type of test meal will always be administered throughout five consecutive days. In total each participant will receive 60 rice meals each meal consisting of approximately 50 g regular unfortified rice, 0.5 g extruded fortified rice, 30 g sauce and 250 ml water. The definite rice amount administered will be decided upon after a pilot investigation. The order of the test meals given in each week will be partially randomized. Thus, if test meals A, B or C will be given throughout 1 week between weeks 1 and 3, test meals D, E and R will be given between weeks 6 and 8. Meals containing iron with the same molecular weight (58 Fe, 57Fe and 54Fe) have to be administered at least 16 days apart from each other, which is the only restriction for randomization. The participants are not allowed to eat after 8 PM and to drink after 12 AM on the day before each study visit, between the meals and for three hours after they finished their second meal, unless they are given snacks by the investigators and are explicitly allowed to eat those. Each meal administration will take approximately 25 minutes. This procedure will be followed for six weeks, with a two weeks break between weeks 3 and 6 (no dietary restrictions within the break-period).

The test meals will be based on 50 g regular unfortified rice and 0.5 g extruded fortified rice (dry weight). The meals will be administered with one of two traditional sauces, with a low (sauce A) or moderate (sauce B) phytic acid (PA) content. Sauce A will be based on tomatoes and onions, sauce B will be based on cowpeas. The rice meals will be prepared individually for each subject, the sauce will be prepared in bulk before the study start. All meals will be served with 250 ml water. The test meals are designed to match ~2/3 of the average dietary requirements in that age-group. In case the rice meals do not provide enough energy (~700 - 900 kcal), the investigators will administer a standardized snack to be consumed during the fasting periods.

ELIGIBILITY:
Inclusion Criteria:

* Iron deficient and/or anemic as per definition;
* Read and signed informed consent form by the caregiver (or has been read out to the caregiver in case of illiteracy);
* Absence of any metabolic-, gastrointestinal or chronic diseases.

Exclusion Criteria:

* Severe underweight (Z-score weight-for-age <-3);
* Severe wasting (Z-score weight-for-height<-3);
* Chronic or acute illness or other conditions that in the opinion of the Principle Investigator (PI) or co-researchers would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol;
* Participants taking part in other studies requiring the drawing of blood;
* Participants who will not be able to comply with the protocol (e.g. plan to move, planned absence, etc.);
* Regular intake (>2 days) of iron-containing mineral and vitamin supplements within the last 2 months.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption | baseline, 6 weeks, 11 weeks
  Change from baseline in the isotopic ratio of iron in blood at week 6 and 11after the administration of test meal including iron isotopes.

SECONDARY OUTCOMES:
Hemoglobin | Baseline, Week 6, Week 11
  Measurements from blood will be given in mg/l.
Plasma Ferritin | Baseline, Week 6, Week 11
  Measurements from blood will be given in mg/l.
C-reactive protein | Baseline, Week 6, Week 11
  Measurements from blood will be given in mg/l.
Zinc protoporphyrin measurement as zinc to heme ratio | Baseline, Week 6, Week 11
Soluble Transferrin receptor in mg/l | Baseline, Week 6, Week 11
Alpha amino glycoprotein in mg/l | Baseline, Week 6, Week 11

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Prof. Dr., Principal Investigator — Swiss FIT
Locations (2):
- University for Development Sciences, Tamale, Northern Region, Ghana
- Swiss Federal Institute of Technology (ETH), Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No